CLINICAL TRIAL: NCT04550169
Title: Evaluation of an Intensive Care Coordination Program to Reduce Use of Hospital Emergency Department Services by Wisconsin Medicaid Members
Brief Title: Wisconsin Evaluation of Emergency Department Care Coordination
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1211; MSN240705 (Other Grant/Funding Number: DHHS, CENTERS FOR MEDICARE & MEDICAID SE); A538500 (Other: UW Madison); SMPH/POP HEALTH SCI/POP HEALTH (Other: UW Madison); Protocol Version April 2020 (Other: UW Madison)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Emergency Department Visit
Keywords: Medicaid; CARES (Wisconsin Client Assistance for Re-Employment and Economic Support)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive Care Coordination: Intensive Care Coordination along with Standard of Care
  Interventions: Other: Intensive Care Coordination
- Control: Standard of Care alone

INTERVENTIONS:
Other: Intensive Care Coordination — Intensive care coordination will include:
  * Discharge instructions and contacts for following up on care and treatment
  * Referral information
  * Appointment scheduling
  * Medication instructions
  * Intensive care coordination by a social worker, case manager, nurse, or care coordinator to connect Medical Assistance (MA) recipient to a primary care provider or to a managed care organization
  * Information about other health and social resources, such as transportation and housing
  * Sharing of information (discharge instructions, medication information, and care plan information) with managed care organization in which patients are enrolled, if applicable
  Groups: Intensive Care Coordination

SUMMARY:
The State of Wisconsin is now expanding its investment in care coordination models as an effort to reduce inappropriate hospital emergency department (ED) use, improve health outcomes, and reduce Medicaid expenditures. This effort begins with a pilot program to support emergency department care coordination in hospitals and health systems that apply and are selected to participate in the pilot program.

The Wisconsin Medicaid program seeks to understand whether this program achieves its intended goals and, specifically, whether the Medicaid payment for such care coordination services produces the intended program outcomes. Hospitals will select members that will receive care coordination services. In a quasi-experimental approach, the study team will compare members that do vs. do not receive the services will be used examine the effects of care coordination and referrals on total ED visits, primary-care treatable ED visits, non-emergent ED visits, and health care costs, as well as the specific effects of referring patients to providers who offer low-cost and after-hours care. To assess the importance of targeting, study team will conduct stratified analyses of vulnerable groups such as people with disabilities and individuals with specific clinical needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are Medicaid enrolled
* Have had 5+ emergency department visits in the past year

Exclusion Criteria:

* Participants who are concurrently eligible for Medicare
* Children (individuals age <18 years).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion Criteria:
  * Adults who are Medicaid enrolled
  * Have had 5+ emergency department visits in the past year
  Exclusion Criteria:
  * Participants who are concurrently eligible for Medicare
  * Children (individuals age <18 years).
Sampling Method: Non-Probability Sample
Enrollment: 3405 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Total Number of Emergency Department Visits | 6 months
Total Number of Emergency Department Visits | 12 months
Total Number of Emergency Department Visits | 18 months
Total Number of Emergency Department Visits | 24 months
Total Number of Emergency Department Visits for Primary Care Preventable and/or Non-Emergent Conditions | 6 months
Total Number of Emergency Department Visits for Primary Care Preventable and/or Non-Emergent Conditions | 12 months
Total Number of Emergency Department Visits for Primary Care Preventable and/or Non-Emergent Conditions | 18 months
Total Number of Emergency Department Visits for Primary Care Preventable and/or Non-Emergent Conditions | 24 months
Cost to Medicaid for all Emergency Department Visits | 6 months
Cost to Medicaid for all Emergency Department Visits | 12 months
Cost to Medicaid for all Emergency Department Visits | 18 months
Cost to Medicaid for all Emergency Department Visits | 24 months
Cost to Medicaid for Emergency Department Use for Primary Care Preventable and/or Non-Emergent Conditions | 6 months
Cost to Medicaid for Emergency Department Use for Primary Care Preventable and/or Non-Emergent Conditions | 12 months
Cost to Medicaid for Emergency Department Use for Primary Care Preventable and/or Non-Emergent Conditions | 18 months
Cost to Medicaid for Emergency Department Use for Primary Care Preventable and/or Non-Emergent Conditions | 24 months

SECONDARY OUTCOMES:
Total Number of Primary Care Visits | 6, 12, 18, and 24 months
Number of Participants Who Used Any Primary Care Visits | 6, 12, 18, and 24 months
Number of Participants Who Used Specialty Care Visits | 6, 12, 18, and 24 months
Total Number of Specialty Care Visits | 6, 12, 18, and 24 months
Number of Participants with Any Hospitalizations | 6, 12, 18, and 24 months
Number of Hospitalization Events | 6, 12, 18, and 24 months
Number of visits to use behavioral health resources, if applicable for the participant | 6, 12, 18, and 24 months
Number of visits to use alcohol and other drug abuse resources if applicable for the participant | 6, 12, 18, and 24 months
Total Cost Related to the Use of Behavioral Health Resources if applicable for the participant | 6, 12, 18, and 24 months
Total Cost Related to Use of Alcohol and other Drug Abuse Resources if applicable for the participant | 6, 12, 18, and 24 months
Total costs of care to Medicaid | 6, 12, 18, and 24 months
Number of participants enrolled in Temporary Assistance for Needy Families (TANF) | 6, 12, 18, and 24 months
Number of participants enrolled in FoodShare | 6, 12, 18, and 24 months
  FoodShare is a program that helps people with limited resources buy the food they need for good health.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Myerson, MPH, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - ThedaCare, Appleton, Wisconsin
  - Ascension Wisconsin, Glendale, Wisconsin
  - Aurora Health Care, Milwaukee, Wisconsin
  - Froedtert Health , Wisconsin, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No